CLINICAL TRIAL: NCT00753792
Title: Multicenter, Randomized, Double Blind, Clinical Trial to Compare the Clinical and Radiological Efficacy of Equivalent Doses of Methylprednisolone Administered Orally or Intravenously in Patients With Multiple Sclerosis During Relapse
Brief Title: Oral Corticotherapy in Megadoses to Treat Multiple Sclerosis During Relapse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Cristina Ramo. MD, Germans Trias i Pujol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CORTEM; 2007-000888-15
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; relapse; methylprednisolone
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): methylprednisolone 1.000 mg/day intravenous administration during three days + placebo of methylprednisolone orally administered
  Interventions: Drug: methylprednisolone; Drug: Placebo
- 2 (Experimental): methylprednisolone 1.250 mg/day orally administered during three days + placebo of methylprednisolone intravenous administered
  Interventions: Drug: methylprednisolone; Drug: Placebo

INTERVENTIONS:
Drug: methylprednisolone — methylprednisolone 1.000 mg/day intravenous administration during three days
  Other Names: Group A
  Arms: 1
Drug: methylprednisolone — methylprednisolone 1.250 mg/day orally administered during three days
  Other Names: Group B
  Arms: 2
Drug: Placebo — Placebo of methylprednisolone administered intravenously (Arm 2) or orally (Arm 1)
  Other Names: Group A; Group B

SUMMARY:
This is a phase IV, multicenter, randomized, double blind clinical trial. The investigators will study 48 patients with remitting relapsing multiple sclerosis (MS) experiencing moderate or severe attack receiving immunomodulatory therapy or not. Patients will be randomly assigned to one of the two groups.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double blind clinical trial to test whether oral methylprednisolone (MP) is not inferior to intravenous methylprednisolone for the treatment of multiple sclerosis (MS) relapse in terms of clinical and radiological efficacy.

Patients will be randomly assigned to one of the following two groups.

Group A: methylprednisolone 1.000 mg/day intravenous administered during three days + placebo of methylprednisolone orally administered

Group B: methylprednisolone 1.250 mg/day orally administered during three days + placebo of methylprednisolone intravenously administered.

Clinical visits will be conducted at 7, 28 and 90 days after treatment starting.

ELIGIBILITY:
Inclusion Criteria:

1. To have been diagnosed MS Remittent Recurrent according to Mc Donald 20052 criteria.
2. To have an EDSS between 0 and 5 before the relapse.
3. The symptoms have begun after at least one month of previous stability.
4. The symptoms have started maximum 15 days before the inclusion.
5. The patient is capable of having an adequate communication with the investigator and to carry out with the clinical trial requisites.
6. To be or not to be with allowed immunomodulatory therapy (IFN-B /AG).
7. To be capable and to be willing to ingest the medication.

Exclusion Criteria:

1. First inflammatory neurological episode (relapse).
2. Multiple sclerosis secondary progressive or primary progressive.
3. The symptoms have gone on for less than 24 hours.
4. To be in treatment or have been treated with corticoids during the three months before.
5. Patients in treatment with immunosuppressors (azathioprine, mitoxantrone, ciclofosfamide...)
6. Pregnancy or breastfeeding or women in fertile age who don't use contraceptives measurements.
7. Illnesses with contraindication treatment with corticoids.
8. Antecedents of serious adverse effects or hypersensitive to related study medication.
9. Patients who wouldn´t be able to perform periodic RMN explorations, patients who are not collaborative or who need anesthesia.
10. Patients with intolerance to lactose.
11. Patients with allergy to contrast used in RMN.
12. Patients with chronic kidney disease.
13. Patients in treatment with natalizumab.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Change in the punctuation of diana functional system score corresponding to in relapse of optic neuritis, trunk's syndrome and myelitis | day 28
Change in EDSS in patients who present a relapse from different type or unknown topography | day 28

SECONDARY OUTCOMES:
Change in the punctuation in each group | between days 7 and 0
Percentage of patients who improve, get worse and keep stable | days 7 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ramo, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (7):
- Spain (7):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital de Mataró, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital de Figueres, Figueres, Girona
  - Hospital Dr. Trueta, Girona, Girona
  - Hospital Arnau de Vilanova, Lleida, Lleida

REFERENCES:
- [Derived] Ramo-Tello C, Tintore M, Rovira A, Ramio-Torrenta L, Brieva L, Saiz A, Cano A, Carmona O, Hervas JV, Grau-Lopez L. Baseline clinical status as a predictor of methylprednisolone response in multiple sclerosis relapses. Mult Scler. 2016 Jan;22(1):117-21. doi: 10.1177/1352458515590648. Epub 2015 Jun 25. PMID 26540732
- [Derived] Grau-Lopez L, Teniente-Serra A, Tintore M, Rovira A, Ramio-Torrenta L, Brieva L, Saiz A, Cano A, Carmona O, Hervas JV, Martinez-Caceres EM, Ramo-Tello C. Similar biological effect of high-dose oral versus intravenous methylprednisolone in multiple sclerosis relapses. Mult Scler. 2015 Apr;21(5):646-50. doi: 10.1177/1352458514546786. Epub 2014 Aug 21. PMID 25145693
- [Derived] Ramo-Tello C, Grau-Lopez L, Tintore M, Rovira A, Ramio i Torrenta L, Brieva L, Cano A, Carmona O, Saiz A, Torres F, Giner P, Nos C, Massuet A, Montalban X, Martinez-Caceres E, Costa J. A randomized clinical trial of oral versus intravenous methylprednisolone for relapse of MS. Mult Scler. 2014 May;20(6):717-25. doi: 10.1177/1352458513508835. Epub 2013 Oct 21. PMID 24144876